CLINICAL TRIAL: NCT01205997
Title: The Effects of Intrathecal Magnesium and Fentanyl Added to Bupivacaine on Postoperative Analgesic Requirement in Patients Undergoing Lower Limb Orthopedic Surgery
Brief Title: Comparison of Postoperative Analgesic Effect of Intrathecal Magnesium and Fentanyl Added to Bupivacaine in Patients Undergoing Lower Limb Orthopedic Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, marzieh beigom khezri, Qazvin University Of Medical Sciences, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ACTRN12610000757011
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Post Operative Pain
Keywords: magnesium; fentanyl; intrathecal; pain
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Fentanyl; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- fentanyl (Active Comparator): Ninety patients 20-60 yr old American Society of Anesthesiologists ( ASA) physical status I or II, scheduled for femur surgery under spinal anesthesia, were studied in a prospective, double-blinded, randomized way. The patients were randomly allocated to one of three groups of 30 each. The magnesium group (groupM) received bupivacaine 15mg combined with 0.5ml magnesium 10%,The fentanyl group (group F) received bupivacaine 15mg combined with0.5 ml fentanyl[25microgram] and The placebo group (group P) received bupivacaine 15mg combined with 0.5ml distilled water(intrathecally) for each three groups 5 minutes prior to surgery)
  Interventions: Drug: Fentanyl
- placebo (Placebo Comparator): Ninety patients 20-60 yr old American Society of Anesthesiologists ( ASA) physical status I or II, scheduled for femur surgery under spinal anesthesia, were studied in a prospective, double-blinded, randomized way. The patients were randomly allocated to one of three groups of 30 each. The magnesium group (groupM) received bupivacaine 15mg combined with 0.5ml magnesium 10%,The fentanyl group (group F) received bupivacaine 15mg combined with0.5 ml fentanyl[25microgram] and The placebo group (group P) received bupivacaine 15mg combined with 0.5ml distilled water(intrathecally) for each three groups 5 minutes prior to surgery)
  Interventions: Drug: placebo(distilled water)
- magnesium sulphate (Active Comparator): Ninety patients 20-60 yr old American Society of Anesthesiologists ( ASA) physical status I or II, scheduled for femur surgery under spinal anesthesia, were studied in a prospective, double-blinded, randomized way. The patients were randomly allocated to one of three groups of 30 each. The magnesium group (groupM) received bupivacaine 15mg combined with 0.5ml magnesium 10%,The fentanyl group (group F) received bupivacaine 15mg combined with0.5 ml fentanyl[25microgram] and The placebo group (group P) received bupivacaine 15mg combined with 0.5ml distilled water(intrathecally) for each three groups 5 minutes prior to surgery)
  Interventions: Drug: magnesium sulphate

INTERVENTIONS:
Drug: Fentanyl — Ninety patients 20-60 yr old American Society of Anesthesiologists ( ASA) physical status I or II, scheduled for femur surgery under spinal anesthesia, were studied in a prospective, double-blinded, randomized way. The patients were randomly allocated to one of three groups of 30 each. The magnesium group (groupM) received bupivacaine 15mg combined with 0.5ml magnesium 10%,The fentanyl group (group F) received bupivacaine 15mg combined with0.5 ml fentanyl[25microgram] and The placebo group (group P) received bupivacaine 15mg combined with 0.5ml distilled water(intrathecally) for each three groups 5 minutes prior to surgery)
  Arms: fentanyl
Drug: placebo(distilled water) — Ninety patients 20-60 yr old American Society of Anesthesiologists ( ASA) physical status I or II, scheduled for femur surgery under spinal anesthesia, were studied in a prospective, double-blinded, randomized way. The patients were randomly allocated to one of three groups of 30 each. The magnesium group (groupM) received bupivacaine 15mg combined with 0.5ml magnesium 10%,The fentanyl group (group F) received bupivacaine 15mg combined with0.5 ml fentanyl[25microgram] and The placebo group (group P) received bupivacaine 15mg combined with 0.5ml distilled water(intrathecally) for each three groups 5 minutes prior to surgery)
  Arms: placebo
Drug: magnesium sulphate — Ninety patients 20-60 yr old American Society of Anesthesiologists ( ASA) physical status I or II, scheduled for femur surgery under spinal anesthesia, were studied in a prospective, double-blinded, randomized way. The patients were randomly allocated to one of three groups of 30 each. The magnesium group (groupM) received bupivacaine 15mg combined with 0.5ml magnesium 10%,The fentanyl group (group F) received bupivacaine 15mg combined with0.5 ml fentanyl[25microgram] and The placebo group (group P) received bupivacaine 15mg combined with 0.5ml distilled water(intrathecally) for each three groups 5 minutes prior to surgery)
  Arms: magnesium sulphate

SUMMARY:
Magnesium has been suggested that NMDA (N-methyl D-aspartate)receptor antagonists induce preemptive analgesia when administrated before tissue injury , thus decreasing the subsequent sensation of pain.

Following Ethics Committee approval and informed patients consent, Ninety patients 20-60 yr old ASA physical status I or II, scheduled for femur surgery under spinal anesthesia, were studied in a prospective, double-blinded, randomized way. The patients were randomly allocated to one of three groups of 30 each. The magnesium group (groupM) received bupivacaine 15mg combined with 0.5ml magnesium 10%,the fentanyl group (group F) received bupivacaine 15mg combined with0.5 ml fentanyl[25microgram] and the placebo group (group P) received bupivacaine 15mg combined with 0.5ml distilled water intrathecally . Time to first requirement of analgesic supplement, Sensory block onset time, maximum sensory level , onset of motor block, duration of blockade, hemodynamics variables, the incidence of hypotension, ephedrine requirements, bradycardia ,hypoxemia [Saturation of peripheral oxygen (SpO2)<90], postoperative analgesic requirements and Adverse events, such as sedation, dizziness , Pruritus and postoperative nausea and vomiting were recorded. Patients were instructed preoperatively in the use of the verbal rating scale (VRS) from 0 to 10 (0no pain, 10maximum imaginable pain) for pain assessment. If the VRS exceeded four and the patient requested a supplement analgesic, methadon5 mg intravenously , was to be given for post-operative pain relief as needed .

ELIGIBILITY:
Inclusion Criteria:

.patients with American Society of Anesthesiologists(ASA) physical status I and

II, undergoing elective femur surgery

-

Exclusion Criteria:

* significant coexisting disease such as hepato-renal and cardiovascular disease
* any contraindication to regional anesthesia such as local infection or ''''bleeding disorders
* allergy to opioids
* long-term opioid use
* history of chronic pain.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2010-08; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Time to first requirement of analgesic supplement | time to first requirement of analgesic supplement from the time of injection intrathecal anesthetic solution
  analgesic administration was initiated by patient request(verbal rating scale[ VRS]>4)
postoperative analgesic requirements | 12 hours postoperative
  postoperative analgesic requirements will be assessed by verbal rating scale (VRS) from 0 to 10 (0no pain, 10maximum imaginable pain).Each administration was initiated by patient request( VRS>4)

SECONDARY OUTCOMES:
Sensory block onset time will be assessed by a pinprick test | sensory block will be assessed by pinprick test every 10 seconds following intrathecal injection
  The onset of sensory block was defined as the time between the end of injection of the intrathecal anesthetic and the absence of pain at the T10 dermatome
duration of sensory block will be assessed by a pinprick test | sensory block will be assessed by pinprick test every 5 minuts following intrathecal injection
  The duration of sensory block was defined as the time between the end of injection of the intrathecal anestheticthe time and regression of two segments from the maximum block height
the onset of motor block will be assessed by the modified Bromage score | every10 seconds following intrathecal injection
  The onset of motor block was defined as the time between the end of injection of the intrathecal anesthetic to Bromage block 1
duration of motor block will be assessed by the modified Bromage score | every 5 minuts following intrathecal injection
  duration of motor block was defined the time from intrathecal injection to Bromage score0
hemodynamic variables is assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 5min before the intrathecal injection
hemodynamic variables is assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 2minutes after intrathecal injection
hemodynamic variables is assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 4minutes after intrathecal injection
hemodynamic variables is assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 6minutes after intrathecal injection
hemodynamic variables is assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 8minutes after intrathecal injection
hemodynamic variables is assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 10minutes after intrathecal injection
hemodynamic variables is assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 15minutes after intrathecal injection
hemodynamic variables is assessed by noninvasive automatic blood pressure measurement and electrocardiogram monitoring | 20minutes after intrathecal injection

CONTACTS AND LOCATIONS:
Overall Officials: Marzieh Beigom Khezri, assistant professor, Principal Investigator — Qazvin medical science university
Locations (1):
- Qazvin university of medical science, Qazvin, Qazvin Province, Iran